CLINICAL TRIAL: NCT00521300
Title: Preoperative Octreotide Treatment of Patients With Growth Hormone Producing Pituitary Adenomas
Brief Title: Preoperative Octreotide Treatment of Acromegaly
Acronym: POTA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-71-98 (REK); S-71-98 (Other: REK); SLKNR 98-5560 (Other: SLK); NCT00241033 (obsolete NCT alias)
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Acromegaly
Keywords: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- octreotide (Experimental): 6 months preoperative treatment with octreotide before transsphenoidal surgery for acromegaly
  Interventions: Drug: Octreotide
- standard surgery (Active Comparator): Standard transphenoidal surgery soon after the diagnosis of acromegaly
  Interventions: Procedure: Direct surgery for acromegaly

INTERVENTIONS:
Drug: Octreotide — First week: Octreotide 50 micrograms subcutaneously three times daily. Second week: Octreotide 100 micrograms subcutaneously three times daily. From the third week on: Octreotide LAR 20 mg intramuscularly every 28th day for 6 months
  Other Names: Sandostatin; Sandostatin LAR
  Arms: octreotide
Procedure: Direct surgery for acromegaly — Direct transsphenoidal surgery
  Arms: standard surgery

SUMMARY:
The purpose of this study is to investigate whether 6 months preoperative treatment with the somatostatin analogue octreotide improves the surgical outcome in patients with acromegaly.

DETAILED DESCRIPTION:
After a baseline evaluation, patients are randomized separately for each study center in blocks of four directly to transsphenoidal surgery or to 6-month preoperative treatment with octreotide.

To reduce the risk of gastrointestinal adverse effects in the pretreatment group, octreotide is initiated at a dose of 50 µg sc three times a day for the 1st week and 100 µg sc three times a day for the 2nd week. From the 3rd week on, the patients receive octreotide LAR (Novartis International AG, Basel, Switzerland) 20 mg im every 28th day for 6 months. Patients receive transsphenoidal surgery within 28 d of the last injection. If surgery are delayed, an extra octreotide LAR injection is given before surgery.

ELIGIBILITY:
Inclusion Criteria:

* GH nadir during a standard 75 g OGTT >= 5.0 mmol/L.
* Pituitary tumor by MRI-scan.

Exclusion Criteria:

* Immediate surgery indicated by usual clinical criteria.
* Pregnant.
* Known adverse effects of octreotide.
* Unfit for participation by any other reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 1999-09; Primary Completion 2005-06 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Surgical cure by transsphenoidal surgery | Primarily 3 months postoperatively, but up to 10 years postoperatively

SECONDARY OUTCOMES:
Effect of treatment on surgical complications and duration of hospital stay, pituitary function, quality of life, and the need for postsurgical medical treatment of acromegaly | Primarily 3 months postoperatively, but up to 10 years postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Sven M Carlsen, MD, PhD, Principal Investigator — Department of Endocrinology, St. Olavs Hospital, University Hospital of Trondheim, Trondheim, Norway
Locations (5):
- Norway (5):
  - Endocrinology Unit, Department of Medicine, Haukeland University Hospital, Bergen
  - Endocrinology Unit, Department of Medicine, Aker University Hospital, Oslo
  - Endocrinology Unit, Department of Medicine, Rikshospitalet-Radiumhospitalet Medical Center, Oslo
  - Endocrinology Unit, Department of Medicine, University Hospital of North Norway, Tromsø
  - Department of Endocrinology, St. Olavs Hospital, Trondheim

REFERENCES:
- [Result] Carlsen SM, Lund-Johansen M, Schreiner T, Aanderud S, Johannesen O, Svartberg J, Cooper JG, Hald JK, Fougner SL, Bollerslev J; Preoperative Octreotide Treatment of Acromegaly study group. Preoperative octreotide treatment in newly diagnosed acromegalic patients with macroadenomas increases cure short-term postoperative rates: a prospective, randomized trial. J Clin Endocrinol Metab. 2008 Aug;93(8):2984-90. doi: 10.1210/jc.2008-0315. Epub 2008 May 20. PMID 18492760
- [Result] Carlsen SM, Svartberg J, Schreiner T, Aanderud S, Johannesen O, Skeie S, Lund-Johansen M, Fougner SL, Bollerslev J; POTA study group. Six-month preoperative octreotide treatment in unselected, de novo patients with acromegaly: effect on biochemistry, tumour volume, and postoperative cure. Clin Endocrinol (Oxf). 2011 Jun;74(6):736-43. doi: 10.1111/j.1365-2265.2011.03982.x. PMID 21521254
- [Result] Fougner SL, Bollerslev J, Svartberg J, Oksnes M, Cooper J, Carlsen SM. Preoperative octreotide treatment of acromegaly: long-term results of a randomised controlled trial. Eur J Endocrinol. 2014 Aug;171(2):229-35. doi: 10.1530/EJE-14-0249. Epub 2014 May 27. PMID 24866574
- [Derived] Olarescu NC, Ueland T, Godang K, Lindberg-Larsen R, Jorgensen JO, Bollerslev J. Inflammatory adipokines contribute to insulin resistance in active acromegaly and respond differently to different treatment modalities. Eur J Endocrinol. 2013 Nov 22;170(1):39-48. doi: 10.1530/EJE-13-0523. Print 2014 Jan. PMID 24092547